CLINICAL TRIAL: NCT07406711
Title: Randomized Controlled Trial on the Effectiveness of a Multidisciplinary Biopsychosocial Program vs Multimodal Treatment in Patients With Chronic Low Back Pain
Brief Title: Biopsychosocial vs Multimodal Chronic Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osijek University Hospital (Other)
Collaborators: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Dijana Hnatesen, Principal Investigator, Osijek University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC-HOSP-R1-14812-2-2021
Record Dates: First submitted 2026-02-01; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Low Back Pain; Multidisciplinary Biopsychosocial Program; Quality of Life
Keywords: chronic low back pain; Multidisciplinary Biopsychosocial Program; Multimodal Treatment; Quality of Life
MeSH Terms: interventions — Physical Therapy Modalities; Combined Modality Therapy; Ultrasonic Therapy; Magnetic Field Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidisciplinary Biopsychosocial Program (Experimental)
  Interventions: Behavioral: Four-week program including group and individual therapy with a multidisciplinary team.Sessions included educational lectures, physical therapy, and multimodal interventions.
- Multimodal Treatment (Active Comparator)
  Interventions: Other: Multimodal treatment. Four-week program including: TENS; Therapeutic ultrasound; Magnetotherapy; Acupuncture. Participants continued their usual prescribed medications.

INTERVENTIONS:
Behavioral: Four-week program including group and individual therapy with a multidisciplinary team.Sessions included educational lectures, physical therapy, and multimodal interventions. — Multidisciplinary Biopsychosocial Program A structured four-week multidisciplinary biopsychosocial treatment program combining patient education, supervised exercise, and individualized care delivered by a multidisciplinary healthcare team. The program addressed physical, psychological, and social aspects of chronic low back pain and included adjunct physical therapy modalities and acupuncture as part of routine clinical care. Participants continued their usual prescribed medications throughout the study.
  Arms: Multidisciplinary Biopsychosocial Program
Other: Multimodal treatment. Four-week program including: TENS; Therapeutic ultrasound; Magnetotherapy; Acupuncture. Participants continued their usual prescribed medications. — Multimodal treatment consisting of physical therapy modalities provided according to standard clinical practice, and acupuncture. Treatment was individualized based on patient needs and did not include a structured multidisciplinary biopsychosocial program. Participants continued their usual prescribed medications throughout the study.
  Arms: Multimodal Treatment

SUMMARY:
This study evaluated the effects of a multidisciplinary biopsychosocial program compared with standard multimodal care in patients with chronic low back pain treated at the University Hospital Osijek. Outcomes included pain intensity, disability, health-related quality of life, anxiety, depression, stress, and sleep quality. Data were collected using standardized self-assessment questionnaires and objective monitoring of sleep and physical activity during a four-week intervention period. The study was conducted as part of a doctoral dissertation.

DETAILED DESCRIPTION:
This prospective, randomized, parallel-group study compared a multidisciplinary biopsychosocial treatment program with standard multimodal care in patients with chronic low back pain treated at the Department of Pain Management, University Hospital Osijek.

Participants were randomly assigned to one of two treatment groups using a random number generator. The multidisciplinary biopsychosocial group participated in a structured four-week program that included patient education, supervised exercise, individualized multidisciplinary care, pharmacotherapy, and acupuncture. The standard multimodal care group received conservative treatment, including pharmacotherapy, physical therapy modalities, and acupuncture.

Clinical and patient-reported outcomes were assessed using standardized self-report questionnaires measuring pain intensity, functional disability, health-related quality of life, anxiety, depression, stress, and sleep quality. In addition, objective data on sleep and physical activity were collected using a wearable smartwatch during the intervention period.

The study was conducted between November 2021 and May 2023 as part of a doctoral dissertation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Chronic low back pain significantly affecting disability and/or emotional distress
* Active use of Croatian language
* Signed informed consent

Exclusion Criteria:

* Age <18 or >65
* Acute pain
* Previous participation in multidisciplinary program
* Pregnancy or cancer-related pain
* Psychotic disorders, moderate-severe cognitive impairment, urgent psychiatric conditions
* PTSD symptoms, extreme fatigue, low motivation, low literacy
* Allergic reactions to metal or silicone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity from baseline to Day 28 measured by Numeric Rating Scale (0-10) | Baseline and Day 28
  Pain intensity is assessed using a self-reported 11-point Numeric Rating Scale (0 = no pain, 10 = worst imaginable pain).
  The outcome represents the change in pain intensity from baseline to Day 28, with greater reductions indicating improvement.

SECONDARY OUTCOMES:
Change in SF-36 Physical Functioning domain score from baseline to Day 28 | Baseline and Day 28
  Health-related quality of life is assessed using the Croatian-validated Short Form-36 questionnaire.
  The outcome represents the change in the Physical Functioning domain score (range 0-100, higher scores indicate better functioning) from baseline to Day 28, with greater increases indicating improvement.
Change in SF-36 Physical Limitations domain score from baseline to Day 28 | Baseline and Day 28
  Health-related quality of life is assessed using the Croatian-validated Short Form-36 questionnaire.
  The outcome represents the change in the Physical Limitations domain score (range 0-100, higher scores indicate fewer physical limitations) from baseline to Day 28, with greater increases indicating improvement.
Change in SF-36 Emotional Limitations domain score from baseline to Day 28 | Baseline and Day 28
  Health-related quality of life is assessed using the Croatian-validated Short Form-36 questionnaire.
  The outcome represents the change in the Emotional Limitations domain score (range 0-100, higher scores indicate fewer emotional limitations) from baseline to Day 28, with greater increases indicating improvement.
Change in SF-36 Energy and Vitality domain score from baseline to Day 28 | Baseline and Day 28
  Health-related quality of life is assessed using the Croatian-validated Short Form-36 questionnaire.
  The outcome represents the change in the Energy and Vitality domain score (range 0-100, higher scores indicate greater energy and vitality) from baseline to Day 28, with greater increases indicating improvement.
Change in SF-36 Psychological Health domain score from baseline to Day 28 | Baseline and Day 28
  Health-related quality of life is assessed using the Croatian-validated Short Form-36 questionnaire.
  The outcome represents the change in the Psychological Health domain score (range 0-100, higher scores indicate better psychological well-being) from baseline to Day 28, with greater increases indicating improvement.
Change in SF-36 Social Functioning domain score from baseline to Day 28 | Baseline and Day 28
  Health-related quality of life is assessed using the Croatian-validated Short Form-36 questionnaire.
  The outcome represents the change in the Social Functioning domain score (range 0-100, higher scores indicate better social functioning) from baseline to Day 28, with greater increases indicating improvement.
Change in SF-36 Physical Pain domain score from baseline to Day 28 | Baseline and Day 28
  Health-related quality of life is assessed using the Croatian-validated Short Form-36 questionnaire.
  The outcome represents the change in the Physical Pain domain score (range 0-100, higher scores indicate less pain) from baseline to Day 28, with greater increases indicating improvement.
Change in SF-36 General Health domain score from baseline to Day 28 | Baseline and Day 28
  Health-related quality of life is assessed using the Croatian-validated Short Form-36 questionnaire.
  The outcome represents the change in the General Health domain score (range 0-100, higher scores indicate better perceived health) from baseline to Day 28, with greater increases indicating improvement.
Change in Oswestry Disability Index (ODI) 2.1a total score from baseline to Day 28 | Baseline and Day 28
  Disability related to low back pain is assessed using the Croatian-validated version of the Oswestry Disability Index (ODI) 2.1a questionnaire.
  The outcome represents the change in the total ODI score (range 0-100, higher scores indicate greater disability) from baseline to Day 28, with greater decreases indicating improvement.
Change in Depression score from baseline to Day 28 measured by the Depression Anxiety Stress Scales-21 (DASS-21) | Baseline and Day 28
  Symptoms of depression are assessed using the Croatian-validated version of the Depression Anxiety Stress Scales-21 (DASS-21).
  The outcome represents the change in the Depression subscale score (higher scores indicate more severe depressive symptoms) from baseline to Day 28, with greater decreases indicating improvement.
Change in Anxiety score from baseline to Day 28 measured by the Depression Anxiety Stress Scales-21 (DASS-21) | Baseline and Day 28
  Symptoms of anxiety are assessed using the Croatian-validated version of the Depression Anxiety Stress Scales-21 (DASS-21).
  The outcome represents the change in the Anxiety subscale score (higher scores indicate more severe anxiety symptoms) from baseline to Day 28, with greater decreases indicating improvement.
Change in Stress score from baseline to Day 28 measured by the Depression Anxiety Stress Scales-21 (DASS-21) | Baseline and Day 28
  Stress symptoms are assessed using the Croatian-validated version of the Depression Anxiety Stress Scales-21 (DASS-21).
  The outcome represents the change in the Stress subscale score (higher scores indicate more severe stress symptoms) from baseline to Day 28, with greater decreases indicating improvement.
Change in Subjective Sleep Quality score from baseline to Day 28 measured by the Pittsburgh Sleep Quality Index (PSQI) | Baseline and Day 28
  Sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI). The outcome represents the change in the Subjective Sleep Quality component score (higher scores indicate worse sleep quality) from baseline to Day 28, with greater decreases indicating improvement.
Change in Sleep Latency score from baseline to Day 28 measured by the Pittsburgh Sleep Quality Index (PSQI) | Baseline and Day 28
  Sleep latency is assessed using the PSQI. The outcome represents the change in the Sleep Latency component score (higher scores indicate longer time to fall asleep and worse sleep) from baseline to Day 28, with greater decreases indicating improvement.
Change in Sleep Duration score from baseline to Day 28 measured by the Pittsburgh Sleep Quality Index (PSQI) | Baseline and Day 28
  Sleep duration is assessed using the PSQI. The outcome represents the change in the Sleep Duration component score (higher scores indicate shorter sleep duration and worse sleep) from baseline to Day 28, with greater decreases indicating improvement.
Change in Habitual Sleep Efficiency score from baseline to Day 28 measured by the Pittsburgh Sleep Quality Index (PSQI) | Baseline and Day 28
  Habitual Sleep Efficiency is assessed using the PSQI. The outcome represents the change in the Habitual Sleep Efficiency component score (higher scores indicate lower sleep efficiency and worse sleep) from baseline to Day 28, with greater decreases indicating improvement.
Change in Sleep Disturbances score from baseline to Day 28 measured by the Pittsburgh Sleep Quality Index (PSQI) | Baseline and Day 28
  Sleep Disturbances are assessed using the PSQI. The outcome represents the change in the Sleep Disturbances component score (higher scores indicate more frequent disturbances and worse sleep) from baseline to Day 28, with greater decreases indicating improvement.
Change in Use of Sleeping Medication score from baseline to Day 28 measured by the Pittsburgh Sleep Quality Index (PSQI) | Baseline and Day 28
  Use of Sleeping Medication is assessed using the PSQI. The outcome represents the change in the Use of Sleeping Medication component score (higher scores indicate more frequent medication use) from baseline to Day 28, with greater decreases indicating improvement.
Change in Daytime Dysfunction score from baseline to Day 28 measured by the Pittsburgh Sleep Quality Index (PSQI) | Baseline and Day 28
  Daytime Dysfunction is assessed using the PSQI. The outcome represents the change in the Daytime Dysfunction component score (higher scores indicate greater daytime impairment) from baseline to Day 28, with greater decreases indicating improvement.
Physical activity / step count measured by Fitbit Charge 3 during the 4-week treatment period | During the 4-week treatment period
  Physical activity / step count is measured using the Fitbit Charge 3 wearable device.
  The outcome represents physical activity / step count summarized across the 4-week treatment period, with higher values indicating greater physical activity.
Sleep quality (Sleep Score) measured by Fitbit Charge 3 during the 4-week treatment period | During the 4-week treatment period
  Sleep quality (Sleep Score) is measured using the Sleep Score generated from sleep stage tracking recorded by the Fitbit Charge 3 wearable device.
  The outcome represents the Sleep Score summarized across the 4-week treatment period, with higher scores indicating better sleep quality.
Change in Pain Catastrophizing Scale (PCS) Rumination subscale score from baseline to Day 28 | Baseline and Day 28
  Pain rumination is assessed using the Rumination subscale of the Pain Catastrophizing Scale (PCS), a validated self-report questionnaire measuring repetitive negative focus on pain.
  The outcome represents the change in the PCS Rumination subscale score from baseline to Day 28, with higher scores indicating greater rumination and greater decreases indicating improvement.
Change in Pain Catastrophizing Scale (PCS) Magnification subscale score from baseline to Day 28 | Baseline and Day 28
  Change in Pain Catastrophizing Scale (PCS) Magnification subscale score from baseline to Day 28
Change in Pain Catastrophizing Scale (PCS) Helplessness subscale score from baseline to Day 28 | Baseline and Day 28
  Pain-related helplessness is assessed using the Helplessness subscale of the Pain Catastrophizing Scale (PCS), a validated self-report questionnaire measuring perceived inability to cope with pain.
  The outcome represents the change in the PCS Helplessness subscale score from baseline to Day 28, with higher scores indicating greater helplessness and greater decreases indicating improvement.
Change in Pain Catastrophizing Scale (PCS) total score from baseline to Day 28 | Baseline and Day 28
  Pain catastrophizing is assessed using the total score of the Pain Catastrophizing Scale (PCS), a validated self-report questionnaire measuring rumination, magnification, and helplessness related to pain.
  The outcome represents the change in the PCS total score from baseline to Day 28, with higher scores indicating greater pain catastrophizing and greater decreases indicating improvement.
Change in painDETECT questionnaire total score from baseline to Day 28 | Baseline and Day 28
  Neuropathic pain features are assessed using the painDETECT questionnaire, a validated self-report screening instrument designed to identify neuropathic pain components. The outcome represents the change in the painDETECT total score from baseline to Day 28, with higher scores indicating a greater likelihood of neuropathic pain and greater decreases indicating improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis AB. Life insurance and the physical examination: a chapter in the rise of American medical technology. Bull Hist Med. 1981 Fall;55(3):392-406. No abstract available. PMID 7037084
- [Background] Tagliaferri SD, Miller CT, Owen PJ, Mitchell UH, Brisby H, Fitzgibbon B, Masse-Alarie H, Van Oosterwijck J, Belavy DL. Domains of Chronic Low Back Pain and Assessing Treatment Effectiveness: A Clinical Perspective. Pain Pract. 2020 Feb;20(2):211-225. doi: 10.1111/papr.12846. Epub 2019 Nov 11. PMID 31610090
- [Background] Skarpsno ES, Mork PJ, Nilsen TIL, Nordstoga AL. Influence of sleep problems and co-occurring musculoskeletal pain on long-term prognosis of chronic low back pain: the HUNT Study. J Epidemiol Community Health. 2020 Mar;74(3):283-289. doi: 10.1136/jech-2019-212734. Epub 2019 Dec 4. PMID 31801790
- [Background] Sirbu E, Onofrei RR, Szasz S, Susan M. Predictors of disability in patients with chronic low back pain. Arch Med Sci. 2020 Jul 8;19(1):94-100. doi: 10.5114/aoms.2020.97057. eCollection 2023. PMID 36817655
- [Background] Hnatesen D, Pavic R, Rados I, Dimitrijevic I, Budrovac D, Cebohin M, Gusar I. Quality of Life and Mental Distress in Patients with Chronic Low Back Pain: A Cross-Sectional Study. Int J Environ Res Public Health. 2022 Aug 26;19(17):10657. doi: 10.3390/ijerph191710657. PMID 36078372
- [Background] Vartiainen P, Heiskanen T, Sintonen H, Roine RP, Kalso E. Health-related quality of life change in patients treated at a multidisciplinary pain clinic. Eur J Pain. 2019 Aug;23(7):1318-1328. doi: 10.1002/ejp.1398. Epub 2019 May 3. PMID 30980782
- [Background] Rivano Fischer M, Persson EB, Stalnacke BM, Schult ML, Lofgren M. Return to work after interdisciplinary pain rehabilitation: One- and two-year follow-up based on the Swedish Quality Registry for Pain rehabilitation. J Rehabil Med. 2019 Apr 1;51(4):281-289. doi: 10.2340/16501977-2544. PMID 30847496
- [Background] Zhang Q, Jiang S, Young L, Li F. The Effectiveness of Group-Based Physiotherapy-Led Behavioral Psychological Interventions on Adults With Chronic Low Back Pain: A Systematic Review and Meta-Analysis. Am J Phys Med Rehabil. 2019 Mar;98(3):215-225. doi: 10.1097/PHM.0000000000001053. PMID 30277912
- [Background] Nielsen A, Dusek JA, Taylor-Swanson L, Tick H. Acupuncture Therapy as an Evidence-Based Nonpharmacologic Strategy for Comprehensive Acute Pain Care: The Academic Consortium Pain Task Force White Paper Update. Pain Med. 2022 Aug 31;23(9):1582-1612. doi: 10.1093/pm/pnac056. PMID 35380733
- [Background] GBD 2021 Low Back Pain Collaborators. Global, regional, and national burden of low back pain, 1990-2020, its attributable risk factors, and projections to 2050: a systematic analysis of the Global Burden of Disease Study 2021. Lancet Rheumatol. 2023 May 22;5(6):e316-e329. doi: 10.1016/S2665-9913(23)00098-X. eCollection 2023 Jun. PMID 37273833
- [Background] Brennan F, Lohman D, Gwyther L. Access to Pain Management as a Human Right. Am J Public Health. 2019 Jan;109(1):61-65. doi: 10.2105/AJPH.2018.304743. PMID 32941757